CLINICAL TRIAL: NCT04623385
Title: Clinical Role of Testosterone and Dihydrotestosterone and Which of Them Should be Inhibited in COVID-19 Patients - A Double-edged Sword?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Faculty of Science, Damietta University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARS -2
Record Dates: First submitted 2020-11-08; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerosolized 13 cis retinoic acid plus Inhalation Inhaled testosterone (Active Comparator): 1. The infected patients will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  2. The infected patients will be treated with a single dose of testosterone (0.1, 0.2, or 0.3 mg) by inhalation for 14 days
  Interventions: Combination Product: Aerosolized 13 cis retinoic acid plus Inhalation Inhaled testosterone
- The standard therapy (Sham Comparator): infected patients will receive the standard therapy for COVID-19 for 14 days
  Interventions: Drug: The standard therapy

INTERVENTIONS:
Combination Product: Aerosolized 13 cis retinoic acid plus Inhalation Inhaled testosterone — 1. The infected patients will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  2. The infected patients will be treated with a single dose of testosterone (0.1, 0.2, or 0.3 mg) by inhalation for 14 days
  Arms: Aerosolized 13 cis retinoic acid plus Inhalation Inhaled testosterone
Drug: The standard therapy — infected patients will receive the standard therapy for COVID-19 for 14 days
  Arms: The standard therapy

SUMMARY:
Clinical Role of Testosterone and Dihydrotestosterone and which of them should be inhibited in COVID-19 patients - A double-edged sword?

COVID-19 attacks and affects Males significantly more than females [1], [2]. Males with COVID-19 are reported to die at twice the rate of females when they come infected with the virus [3]. The upregulation of TMPRSS2 by androgens could explain the increased susceptibility to COVID-19 in men.Contrary to expected, as a study demonstrated that The expression level of TMPRSS2 increased 6-fold in androgen stimulated LNCaP cells, relative to androgen-deprived cells[4]. But, surprisingly, low levels of testosterone led to the over expression and upregulation of ACE2 and TMPRSS2 receptors, facilitating SARS-CoV-1 entry into the alveolar cells, and deregulating a lung-protective pathway [5].According to literature Dihydrotestosterone is many times more potent than testosterone, and many of the effects that testosterone has in the body only happen after it is converted to dihydrotestosterone [6]. Therefore, we hypothesis that testosterone has better effect than dihydrotestosterone in case of COVID-19, because a study found that DHT significantly induced the expression of TMPRSS2 [7]. And at the same time , decreased testosterone levels in critically diseased males harmfully affect pulmonary endothelial cell functioning, impair the ability to clear the virus , promote systemic . Obesity among males, promote defective immune response, , and also generates more pro-inflammatory cytokines important in cell signaling, emanating in increased, severe disease, worst outcome and vulnerability. Insufficient serum testosterone level is a poor prognostic indicator for patients infected with COVID-19 by downregulation pulmonary protective pathways [5], [8]. On the contrary, high testosterone levels can lead to complication of thrombosis which is also one of the serious manifestations in COVID-19 patients[9]. Thereby we hypothesize that decreased testosterone levels in men have a direct relation with the severity of infection and a worse outcome in COVID-19. In this case we should found an appropriate treatment that induces testosterone level to introduce its protective effect and up regulate pulmonary protective pathways and at the same time protect against thrombosis and works to reduce the impact of dihydrotestosterone on lung cells preventing up regulation of TMPRSS2, Her we shed new light on the appropriate treatment can overcome the challenges that face testosterone therapy in the era of COVID-19 After searching MEDLINE , PubMed, , Google Scholar, preprints and Controlled Trials until September , 2020 we found that the appropriate treatment in this case is aerosolized 13 cis retinoic acid in combination with testosterone therapy, as more than one study found that 13 cis retinoic acid reversibly and potentially inhibit the effect of dihydrotestosterone on different targeted cells. In addition its impact on thrombin.

DETAILED DESCRIPTION:
The study is a randomized interventional comparative Phase IIII trial. 1000 adult male and female patients with positive COVID-19 diagnosis and fulfilling the below outlined inclusion criteria will be enrolled into the study.

After searching PubMed, MEDLINE, Google Scholar, preprints and Controlled Trials until September , 2020 we found that the best and appropriate drug which can be combined with testosterone replacement therapy is aerosolized 13 cis retinoic acid owing to its impact on DHT and thrombin in addition it can be given in the form of aerosol for targeting pulmonary cells with minimal systemic side effects . As previous study found that testosterone therapy (TTh) administration using both topical and injectable formulations yielded transient and concomitant rises in both DHT and T, with higher Hct elevations in men with higher DHT and T levels[38]. As Testosterone is converted to DHT by the action of 5 alpha-reductase enzyme at these target tissues.[39]. DHT is a potent activator of TMPRSS2[31,4] and this will be followed by the activation of COVID-2019 spike protein to bind to its ACE2 receptors in lung which in turn makes it more vulnerable to covid-19. A study demonstrated that 13- cis -Retinoic acid competitively and reversibly inhibits dihydrotestosterone.[40] on contrary to other selective inhibitor of serum DHT which led to sexual adverse effects because it usually given systemically which increases the chance of systemic serious side effects . But 13- cis -Retinoic acid will be given in the form of aerosol to avoid these systemic side effects. Therefore, we suggest that 13- cis -Retinoic acid will downregulate TMPRSS2 expression thorough temporary preventing the effect of dihydrotestosterone (DHT) on the activation of TMPRSS2 gene expression. Furthermore, 13- cis -Retinoic acid Found to exert potential effect on thrombin as high testosterone levels can lead to thrombosis which is also one of the fatal manifestations in COVID-19 patients .A study in vitro found that Retinoic acid showed the highest inhibition of both the forms of thrombin [41].

Moreover, we hypothesize that any drug which downregulates TMPRSS2 expression through targeting AR, AR co-regulatory factors, or AR downstream transcription factors might be potentially effective against COVID-19 and is worth investigating under a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

* Hypercholesterolemia
* Hypertriglyceridemia
* Liver disease
* Renal disease
* Sjögren syndrome
* Pregnancy
* Lactation
* Depressive disorder
* Body mass index less than 18 points or higher than 25 points
* Contraindications for hormonal contraception or intrauterine device.
* Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
* Patients receiving anti-hcv treatment
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
* Known malignant disease, PSA > 3 ug/L, Nycturia > 3 times
* The competent physician considered it inappropriate to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7and 14 days
  Proportion of lung injury score decreased or increased after treatment

SECONDARY OUTCOMES:
Absolute lymphocyte counts | at 7and 14 days
  lymphocyte counts
Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon | at 7and 14 days
  Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon
Serum level of COVID19 RNA | at 7and 14 days
  Serum level of COVID19 RNA
Angiotensin 1-7 (Ang 1-7) changes over time | at 7and 14 days
  Angiotensin 1-7 (Ang 1-7) changes over time
Angiotensin 1-5 (Ang 1-5) changes over time | at 7and 14 days
  Angiotensin 1-5 (Ang 1-5) changes over time
Renin changes over time | at 7and 14 days
  Renin changes over time
Aldosterone changes over time | at day 7 and 14
  Aldosterone changes over time
Angiotensin-converting enzyme (ACE) changes over time | at day 7 and 14
  Angiotensin-converting enzyme (ACE) changes over time
Frequency of adverse events and severe adverse events | at day 7 and 14
  Frequency of adverse events and severe adverse events
Transe membrane protease ,serine II (TMPRSS2) changes over time | day 7 and 14
  Transe membrane protease ,serine II (TMPRSS2) changes over time
Testosterone levels changes over time | day 7 and 14
  Testosterone levels changes over time
Dihydrotestosterone(DHT) levels changes over time | day 7 and 14
  Dihydrotestosterone(DHT) levels changes over time
Cholesterol levels changes over time | day 7 and 14
  Cholesterol levels changes over time
Thrombin time (TT) | day 7 and 14
  Thrombin time (TT)